CLINICAL TRIAL: NCT06833593
Title: Efficacy of Optimized Antimicrobial Combination Therapy for Treatment of Enterococcus Faecalis Bacteremia and Identification of Intestinal Microbiota Signature
Brief Title: Antimicrobial Combination Therapy for Treatment of Enterococcus Faecalis Bacteremia
Acronym: MicroEFfAECT
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: Micro-EFfAECT; "Ricerca Finalizzata 2019" (Other Grant/Funding Number: Italian Ministry of Health)
Record Dates: First submitted 2024-12-30; First posted 2025-02-19 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-10

CONDITIONS: Enterococcus Faecalis Infection; Blood Stream Infection; Gut Microbiomes
Keywords: Enterococcus faecalis bloodstream infection; Human tissue analysis in vitro; Gut microbiota analysis; Enterococcus faecalis genomic analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * isolated bacterial strains for genomic analysis
  * stool samples for gut microbiota analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult with Enterococcus faecalis monomicrobial bloodstream infection: Adult patients with primary Enterococcus faecalis monomicrobial bloodstream infection

SUMMARY:
Prospective, multicenter, national, observational pharmacological study on the evaluation of efficacy of appropriate monotherapy vs combination treatment for non-complicated Enterococcus faecalis (EF) bloodstream infection (BSI) and identification of gut microbiota fingerprint of patients with EF-BSI correlated to antimicrobial treatment and clinical outcome

DETAILED DESCRIPTION:
Enterococcus faecalis (EF) is a common commensal of human gastrointestinal tract that can act as opportunistic pathogen causing mild to severe clinical illness. Severe infections due to EF include bacteremia, endocarditis and catheter-related infections. EF is the fourth causative pathogen of bloodstream infection (BSI) in Europe after E. coli, S. aureus and S. pneumoniae. The incidence of infections caused by E. faecalis has increased over the last decades probably as a consequence of the global aging of the population. EF-BSI is associated to a high mortality rate (11-26% of cases).The main factors that may contribute to short-term mortality are the number of comorbidities, the need of admission in intensive care unit and the prompt administration of appropriate antibiotic treatment.

The optimal treatment of EF-BSI uncomplicated with endocarditis is still a matter of debate. Ampicillin is commonly considered the drug of choice, when active in vitro. However, several studies demonstrated the synergistic effect of the combination treatment with an aminoglycosides or ceftriaxone in case of life-threatening infections. To date the efficacy of the combination treatment in patients with EF-BSI was poorly evaluated in clinical studies and most of the data come from very old uncontrolled clinical observations. One strategy for overcoming this uncertainty is to assess the synergistic interaction of different antimicrobial molecules by in vitro tests and to validate in vitro synergisms with clinical studies. Indeed, in vitro evaluation of the drug combination effect has the potentiality for improving treatment by suggesting the possible synergistic or antagonistic interaction of antimicrobial associations. Although, different studies suggested the potential clinical utility of synergy testing, the real prognostic value of these methods is not defined yet. In this context, synergy testing could be used as strategy for improving antibiotic treatment of EF-BSI by suggesting the optimal antimicrobial combination therapy. Ceftaroline and ceftobiprole are two novel cephalosporins, which exhibit intrinsic activity against methicillin-resistant S. aureus. Both drugs seem to show a good level of affinity to penicillin binding protein (PBP) 5, a class B, commonly expressed by Enterococcus spp. The use of these drugs in association with ampicillin or daptomycin seems promising. However, clinical efficacy of these combinations is not well defined yet. Gut microbiota of healthy individual is composed by a consortium of bacteria balanced by symbiotic or antagonistic relationships. Antimicrobial treatments altered this equilibrium conferring competitive advantage for different species, including host pathogens. Disruption of the balance in the gut microbial composition has been associated to different pathological conditions (metabolic disease, type 2 diabetes, colorectal cancer or inflammatory bowel disease). Also, administration of antimicrobials contributes to increase resistome in the intestinal microbiota and diffusion of antimicrobialresistant pathogens through selective pressure. The central objective of this study is to identify the gut microbiota signature associated to different antimicrobial therapy of EF-BSI and to clinically validate novel diagnostic tools for optimizing antimicrobial therapy in critically ill patients.

The primary aim of the study is to compare efficacy of appropriate monotherapy vs combination treatment for EF-BSI and validate clinically the in vitro synergistic/antagonistic interaction of antimicrobial combinations by synergy tests.

Secondary objectives are:

* To define the prognostic and predictive value of EF genotypic and phenotypic traits on the basis of antimicrobial treatment and clinical outcome
* To compare gut microbiota fingerprint of patients with EF-BSI and correlate to antimicrobial treatment and clinical outcome

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years)
* Monomicrobial EF-BSI
* Receipt of ≥ 5 days of at least one in vitro active drug (ampicillin, amoxicillin/clavulanate, ampicillin/sulbactam, piperacillin, vancomycin, teicoplanin, daptomycin and linezolid) with or without a synergistic drug (ceftriaxone, gentamycin, streptomycin), at common suggested dosages for EF-BSI in empirical or definitive therapy
* Written informed consent

Exclusion Criteria:

* Short term (within 3 days from BSI) mortality
* Other concomitant infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients (≥ 18 years) with primary Enterococcus faecalis monomicrobial bloodstream infection
Sampling Method: Non-Probability Sample
Enrollment: 510 (Estimated)
Dates: Start 2021-02-06 (Actual); Primary Completion 2026-09-26 (Estimated); Study Completion 2026-09-26 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Clinical Cure and Improvement Rates for EF-BSI | Up to 6 weeks from patient enrollment, with bacterial strains isolated at baseline
  The clinical cure and improvement rates will be evaluated for patients undergoing mono therapy and combination therapy for EF-BSI.
Comparison of Clinical Outcomes Between Mono Therapy and Combination Therapy | Up to 6 weeks from patient enrollment, with bacterial strains isolated at baseline
  A comparison of clinical outcomes between mono therapy and combination therapy in terms of clinical cure, improvement, and any adverse events.
Validation of In Vitro Synergy Tests | Up to 6 weeks from patient enrollment, with bacterial strains isolated at baseline
  To validate the in vitro synergy or antagonism of antimicrobial combinations tested in the laboratory, correlating these results with clinical outcomes. In vitro synergy tests will be conducted to evaluate the interaction between antimicrobial combinations, and the results of these tests will be correlated with the clinical outcomes of the patients.

SECONDARY OUTCOMES:
Genotypic Analysis of E. faecalis | From enrollment to the end of the follow-up at three months
  To explore how the genotypic (e.g., resistance and virulence genes) and phenotypic traits of E. faecalis strains influence infection severity, antimicrobial treatment response, and clinical outcomes. Define the prognostic and predictive value of these genotypic and phenotypic traits based on antimicrobial treatment and clinical outcomes. Genomic analyses will be conducted to identify antimicrobial resistance determinants, clonal relationships through multilocus sequence typing (MLST), and virulence factor genes for To explore how the genotypic traits (e.g., antimicrobial resistance and virulence genes) of E. faecalis strains influence infection severity, antimicrobial treatment response, and clinical outcomes. Weekly genomic analyses will be conducted to identify antimicrobial resistance determinants, clonal relationships through multilocus sequence typing (MLST), and virulence factor genes for each E. faecalis genome.
Phylogenetic Relationship and Clonal Diversity | From enrollment to the end of the follow-up at three months
  A phylogenetic tree will be constructed based on the core genome of clinical E. faecalis isolates. This will allow the identification of clonal relationships and shared genetic factors among the strains. A deeper genetic analysis will also be performed to explore genetic factors that may influence infection outcomes.
Correlation Between Genotypic/Phenotypic Traits and Clinical Outcome | From enrollment to the end of the follow-up at three months
  The prognostic and predictive value of the genotypic (e.g., resistance and virulence genes) and phenotypic traits of E. faecalis will be defined in relation to antimicrobial treatment and clinical outcomes. A comprehensive E. faecalis genomic database will be created to correlate these traits with infection severity, antimicrobial treatment, and clinical outcomes. The correlation will be explored through weekly genomic analyses and clinical data review.
Gut Microbiota Fingerprint Analysis in EF-BSI Patients | From enrollment to the end of the follow-up at three months
  To compare the gut microbiota fingerprint of patients with E. faecalis bloodstream infections (EF-BSI) and correlate it with antimicrobial treatment and clinical outcomes. Faecal samples will be collected during antimicrobial therapy and 90 days after therapy withdrawal. These samples will be analyzed for 16S rRNA and the relative microbial composition. Clinical conditions, diet, infection relapse after therapy withdrawal, and their correlation with antimicrobial treatment and faecal abundance will also be evaluated.
Intestinal Microbiota Composition and Its Correlation with Treatment Outcomes | From enrollment to the end of the follow-up at three months
  To evaluate the relationship between antimicrobial treatment, gut microbiota composition, and clinical outcomes (such as infection relapse, health status, or disease progression). Faecal samples will be collected from patients with EF-BSI treated with different antimicrobial therapies. These samples will be analyzed for 16S rRNA and relative microbial abundance. The clinical conditions, diet, infection relapse after therapy withdrawal, and their correlation with antimicrobial treatment and faecal abundance will also be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Maddalena Giannella, MD PhD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (4):
- Italy (4):
  - Ospedale Maggiore "Carlo Alberto Pizzardi" di Bologna, Bologna, Bologna
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna
  - Azienda Ospedaliero Universitaria di Catanzaro "Mater Domini", Catanzaro, Catanzaro
  - Humanitas Research Hospital, Milan, Milano